CLINICAL TRIAL: NCT02914574
Title: The Patellofemoral Pain Functional Performance and Arthrogenic Muscle Inhibition Study
Brief Title: The Patellofemoral Pain Functional Performance Study
Acronym: PFP-FP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Henrike Greuel, PhD student, Principal Investigator, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSCR15-143
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Patellofemoral Pain; Anterior Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- healthy control (Other): Healthy control group will attend one visit and functional performance, muscle strength and flexibility, quadriceps AMI, patellar position and posture will be measured. No intervention will be applied.
  Interventions: Other: PowersTM strap

INTERVENTIONS:
Other: PowersTM strap — The powers strap aims to decrease knee varus through supporting femoral abduction and external rotation. Participants will wear the Powers strap while performing functional tasks (running, squatting, single leg step down).

SUMMARY:
This study primarily aims to investigate arthrogenic muscle inhibition (AMI), an underlying mechanism in patellofemoral pain (PFP), which remain to date understudied. Although, studies have revealed that AMI needs to be eliminated before improvements in muscle strength can be achieved, to date quadriceps muscle inhibition in patients with PFP remains understudied. To date the influence of AMI on functional performance and the direct link to pain in patients with PFP remain unclear. This study aims to investigate the link between AMI to pain, functional performance and how an acute treatment can affect functional performance and pain.

DETAILED DESCRIPTION:
Patellofemoral pain (PFP) is one of the most frequently diagnosed conditions in patients with knee complaints.

Studies investigating the therapeutic effect on PFP revealed that the majority of patients with PFP were still suffering of knee pain after 5 to 8 years, despite initially received treatment and education, indicating that the current treatments fail to prevent the chronicity of symptoms. Considering that current treatment-strategies of patients with PFP seem to be unable to avoid the development of chronic symptoms, the question arises if the underlying factors of PFP are understood sufficiently.

In contrary to the current broad body of literature on weakness, potentially underlying factors which might influence or even lead to PFP, such arthrogenic muscle inhibition (AMI) or the break phenomenon remain understudied.

Pain in PFP has been proven to be linked to quadriceps strength deficit, gluteal strength deficits, knee stability, irregularities in the quadriceps torque curve, and functional performance. Bazett et al. (2011) described that pain "is more than a symptom and might play a role in the etiology or progression of PFP". Furthermore, pain seems to play a crucial role in AMI. However, the correlation between pain and AMI in patients with PFP has not been investigated currently.

No assessment in isolation can provide a full picture of the problem. The combination of AMI, the break phenomenon with a biomechanical analysis might enable the determination of the impact of inhibition and strength on biomechanical changes. In addition, it might provide an answer to whether AMI or weakness cause biomechanical alterations, which would help to optimise treatment approaches in PFP.

The PowersTM strap strap was developed with the aim of assisting lower limb kinematics, decreasing knee varus through supporting femoral abduction and external rotation. This treatment may potentially also directly improve functional performance. As the functional performance in participants with PFP after the application of the PowersTM strap has not been investigated, this study aims to analyse if there is a direct link between the application of the PowersTM strap to functional performance and pain.

ELIGIBILITY:
Inclusion Criteria for patients with PFP:

1. Reproducible pain with at least two of these activities: ascending or descending stairs or ramps, squatting, kneeling, prolonged sitting, hopping/ jumping, isometric quadriceps contraction or running
2. Clearly defined pain location in the peripatellar region
3. Reports of pain greater than 1 month duration.
4. They are able to perform squatting, running and MVC task- Participant response
5. Age range: 18-45 years old

Inclusion criteria for healthy volunteers:

1. Healthy and without any previous lower limb injuries
2. The participant is able to perform squatting, running and MVC task

Exclusion Criteria:

1. Previous history of knee surgery
2. Previous history of (traumatic) patella dislocation or instability
3. Previous history of ligamentous instabilities
4. Previous history of traumatic, inflammatory or infectious pathology in the lower extremity
5. Previous history of internal derangement or other causes
6. Previous diagnosed degenerative conditions in the knee
7. Exclusion if patients cannot perform running, step down, or MVC task.
8. Exclusion criteria for the healthy control group are: clinical evidence of other knee injury or knee pain, and current significant injury affecting other lower extremity joints.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Influence of Powers strap | 1 day
  The influence of the Powers strap on functional performance will be investigated by analysing hip and knee kinematics and kinetics with and without the Powers strap in participants with PFP

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salford, Salford, Greater Manchester, United Kingdom